CLINICAL TRIAL: NCT06364150
Title: Therapeutic Use of Angiopoietin-Primed Autologous Peripheral Blood Stem Cell in Myocardial Infarction
Acronym: MAGICcell6
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National Hospital (Other Government)
Collaborators: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hyun-Jai Cho, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MAGIC6
Record Dates: First submitted 2024-03-28; First posted 2024-04-15 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-04

CONDITIONS: Acute Myocardial Infarction
Keywords: Peripheral Blood Stem Cell Treatment; Acute Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: This is a single arm, open label interventional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cell treatment arm (Experimental): Patients who receive Angiopoietin-Primed Autologous Peripheral Blood Stem Cell in Myocardial Infarction
  Interventions: Biological: Autologous Peripheral Blood Stem Cell injection

INTERVENTIONS:
Biological: Autologous Peripheral Blood Stem Cell injection — For peripheral blood stem cell mobilization, G-CSF and EPO will be injected for a total of 4 days, followed by collection of mobPBSC via apheresis. In ex-vivo setting, mobPBSC will be primed with Ang1 for 1 hour. A total of 2 X109 Ang1 primed mobPBSC will be injected to the culprit artery.

SUMMARY:
This study will evaluate the efficacy and safety of "Therapeutic Use of Autologous-Primed Autologous Peripheral Blood Stem Cell Treatment for Myocardial Regeneration in Acute Myocardial Infarction".

DETAILED DESCRIPTION:
Patients diagnosed with acute myocardial infarction will receive percutaneous coronary intervention to the culprit coronary artery according to standard procedures. For peripheral blood stem cell mobilization, Granulocyte colony-stimulating factor (G-CSF) and erythropoietin (EPO) will be injected for a total of 4 days, followed by collection of mobilized peripheral blood stem cell (mobPBSC) via apheresis. In ex-vivo setting, mobPBSC will be primed with angiopoietin 1 (Ang1) for 1 hour. A total of 2 X109 Ang1 primed mobPBSC will be injected to the culprit artery.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male and female aged ≥19 years and ≤ 80 years
* 2. A clinical diagnosis of acute myocardial infarction within 4 weeks from randomization
* 3. Successful percutaneous coronary intervention to the target lesion (TIMI flow grade 3 and residual stenosis <30% at the target lesion) with a drug-eluting stent and/or drug-eluting balloon
* 4. Agreement to give written informed consent.

Exclusion Criteria:

1. Patients with uncontrolled heart failure (Killip class ≥ grade 2, or left ventricular ejection fraction <20%)
2. Patients with uncontrolled chest pain due to ischemia
3. Patients with uncontrolled arrythmia
4. Active malignancy, or incompletely treated malignancy
5. Active infectious disease
6. Uncontrolled hematologic disease, including coagulopathy or bleeding diathesis
7. Presence of non-cardiac comorbidity with life expectancy ≤1 year from randomization
8. Females with childbearing potential or breast-feeding
9. Refusal to give written informed consent
10. Other conditions that may result in protocol non-compliance by the committees

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Left ventricular systolic function | 12 months after treatment
  Left ventricular ejection fraction measured by echocardiography (measured in percent)

SECONDARY OUTCOMES:
Regional wall motion score index | 12 months after treatment
  Regional wall motion score index measured by echocardiography. The score is scaled from 1.0 to 4.0. Using a standard transthoracic echocardiography sequence, each one of the 16 myocardial segments are assigned a score from 1 to 4. The scores for 16 segments are scaled as normokinesia (1 point) or hypokinesia (2 points) or akinesia (3 points) or dyskinesia (4 points). A score of 1.0 is considered normokinetic, and a score of 3.0 correlated as akinetic.
B-natriuretic peptide level | 12 months after treatment
  Laboratory test which is measured in picograms per milliliter (pg/ml).
6-minute walk test | 12 months after treatment
  6-minute walk test is measured in meters.
All-cause death | 12 months after treatment
  Rate of patients with a mortality event due to any cause
Target lesion Revascularization | 12 months after treatment
  Rate of patients who received additional revascularization for the target lesion (the coronary lesion that was treated at the index procedure)
Readmssion | 12 months after treatment
  Rate of patients who were readmitted due to any cause
Cardiovascular death | 12 months after treatment
  Rate of patients with a mortality event due to cardiovascular cause
non-Target lesion Revascularization | 12 months after treatment
  Rate of patients who received additional revascularization for a non-target lesion (the coronary lesion that was NOT treated at the index procedure)

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Jai Cho, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Any request for data sharing should be sent as an inquiry to the principle investigator.